CLINICAL TRIAL: NCT00907049
Title: Study of the Association Between Neck Pain and the Quality of Sleep
Brief Title: Association Between Neck Pain and Quality of Sleep
Status: Completed | Type: Observational
Sponsor: Kovacs Foundation (Other)
Responsible Party: Principal Investigator, Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation, Kovacs Foundation
Other Study IDs: FK-30
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Neck Pain; Disability
Keywords: quality of sleep; neck pain; disability; catastrophizing; depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neck Pain; Depression

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subacute neck pain; chronic neck pain: Patients with subacute or chronic neck pain seen in the Primary Care Centers participating in the study.

SUMMARY:
A prospective study to assess the association between the change in quality of sleep and the change in intensity of pain in Spanish patients seen for subacute or chronic neck pain. The objective is to determine the prevalence of sleep alterations, the association between quality of sleep and intensity of pain, degree of disability, intensity of catastrophizing and depression.

ELIGIBILITY:
Inclusion Criteria:

* patients with nonspecific neck pain of more than 14 days duration
* seen in health centers participating in the study
* patients who accept to participate and sign the consent form
* without age limits and regardless of gender

Exclusion Criteria:

* inability to complete the questionnaires (illiteracy, dementia)
* inflammatory rheumatologic disease, fibromyalgia, cancer in last 5 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen for neck pain in the primary care centers participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2009-09; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the association between neck pain and quality of sleep in patients with subacute or chronic nonspecific neck pain. | 3 months

SECONDARY OUTCOMES:
Assessment of the association between quality of sleep and disability, catastrophizing and depression in patients with subacute or chronic nonspecific neck pain. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Víctor Abraira, PhD, Principal Investigator — Hospital Ramón y Cajal, Unidad de Bioestadística Clínica, Madrid, Spain
Locations (2):
- Spain (2):
  - Kovacs Foundation, Palma de Mallorca, Balearic Islands
  - Hospital Ramón y Cajal, Madrid, Madrid

REFERENCES:
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Moldofsky H. Sleep and pain. Sleep Med Rev. 2001 Oct;5(5):385-396. doi: 10.1053/smrv.2001.0179. PMID 12531004
- [Background] McCracken LM, Iverson GL. Disrupted sleep patterns and daily functioning in patients with chronic pain. Pain Res Manag. 2002 Summer;7(2):75-9. doi: 10.1155/2002/579425. PMID 12185371